CLINICAL TRIAL: NCT04746807
Title: Barriers to Physical Activity in People With MS (Barrieren für körperliche Aktivität Bei MS-Betroffenen - BarKA-MS) - A Longitudinal Observational Study
Brief Title: Barriers to Physical Activity in People With MS
Acronym: BarKA-MS
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Dr. Roman Gonzenbach, Kliniken Valens (Unknown)
Responsible Party: Principal Investigator, Viktor von Wyl, Viktor von Wyl, University of Zurich
Other Study IDs: 1
Record Dates: First submitted 2021-01-28; First posted 2021-02-10 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; physical acitivity; digital mobility measurements; real-life assessments
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multiple Sclerosis (MS) is a chronic inflammatory disease leading to the demyelination of the central nervous system. Promoting physical activity has gathered attention as an effective means to improve health-related quality of life and to mitigate symptoms such as fatigue and depressive symptoms in individuals suffering from MS. However, persons suffering from MS often experience difficulties in staying active. A comprehensive understanding of barriers to staying physical active for persons with MS in Switzerland is currently lacking. Given the importance of physical activity in the context of MS a detailed understanding of this matter would be key for future research and treatment.

A key challenge when studying physical activity in the context of MS is to obtain objective and accurate measurements that are not prone to reporting bias. While accelerometer-based measurements hold promise in this regard they are not convenient for routine implementation in real-world environments. Initial research has identified consumer-grade wearables such as Fitbits as a promising alternative whereby focusing on the main outcome average step count. Given the rich detail of activity patterns that can be derived from such devices, research has so far underutilized the available information that has the potential to provide more comprehensive insight into this matter.

Objectives: The present project aims to determine the common factors in real-life settings limiting physical activity in persons with MS and the impact of these barriers on physical activity. Further, the present study aims to provide precedence for future research investigating physical activity in MS by examining the quality, reliability, internal consistency, and validity of PA metrics derived from the wide-spread consumer-grade activity tracker Fitbit in comparison to an accelerometer.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* definite diagnosis of relapsing or progressive MS (i.e., confirmed by their physician)
* persons with reduced walking ability but who are still able to walk independently with or without an assistive device (e.g., as expressed by an Expanded Disability Status Scale score between 3-6.5)
* possess a personal computer, mobile phone or a tablet with Bluetooth functionality,
* be willing and able to perform study procedures,
* be able to provide informed consent
* be able to answer the questionnaires in German.

Exclusion Criteria:

* serious illnesses that preclude safe participation in physical activity
* inability to follow study procedures
* inability to complete questionnaires in German
* inability to complete baseline questionnaires or activate the Fitbit device will lead to the exclusion of the participant from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A minimum of 30 and maximum of 45 patients will be enrolled in this study. Patients undergoing an inpatient rehabilitation program at Kliniken Valens.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-11-14 (Actual); Study Completion 2021-11-14 (Actual)

PRIMARY OUTCOMES:
Step count (Fitbit) | measured continuously over the course of the study, on average of 7-8 weeks
Step count (Accelerometer) | measured continuously during the last week at rehab stay and first week at home (= 2 weeks in total)
International Physical Activity Questionnaire-Short Form (IPAQ-SF) | Time Frame: change from T0 (baseline), at week 1 - 8 (1 - 8 week after T0)
Perceived Barriers to Physical Activity | Time Frame: change from T0 (entry to study) at post-treatment (2-4 weeks after T0), change from T0 at 4 weeks follow-up (6-8 weeks after T0)
  Perceived Barriers to Physical Activity will be assessed by a modified version of the Barriers to Health Promoting Activities for Disabled Persons Scale. The original version of this instrument lists 18 barriers and asks participants to indicate "how much each of these problems [the barriers] keeps you from participating in health-promoting activities." This scale has been previously modified to measure barriers to physical activity, instead asking participants to indicate "how much each of these problems keeps you from participating in physical activity and exercise".

SECONDARY OUTCOMES:
Health status and Health-Related Quality of Life (EQ-5D-5L) | Time Frame: change from T0 (entry to study) at post-treatment (2-4 weeks after T0), change from T0 at 4 weeks follow-up (6-8 weeks after T0)
Patient Health Questionnaire depression scale (PHQ-8) | Time Frame: change from T0 (entry to study) at post-treatment (2-4 weeks after T0), change from T0 at 4 weeks follow-up (6-8 weeks after T0)
Generalized Self Efficacy Scale (GSE) | Time Frame: change from T0 (entry to study) at post-treatment (2-4 weeks after T0), change from T0 at 4 weeks follow-up (6-8 weeks after T0)
Fatigue Scale for Motor and Cognitive Functions (FSMC) | Time Frame: change from T0 (entry to study) at post-treatment (2-4 weeks after T0), change from T0 at 4 weeks follow-up (6-8 weeks after T0)
Valens in-house pain scale | Time Frame: change from T0 (entry to study) at post-treatment (2-4 weeks after T0), change from T0 at 4 weeks follow-up (6-8 weeks after T0)
  Pain will be assessed using three 11-point scales (0 = no pain at all; 10 = strongest pain I can imagine). Participants will be asked to rate pain intensity at the present moment as well as minimal and maximal pain intensity over the previous week.
MS Walking Scale-12 (MSWS-12) | Time Frame: change from T0 (entry to study) at post-treatment (2-4 weeks after T0), change from T0 at 4 weeks follow-up (6-8 weeks after T0)
Timed Up and Go (TUG) | Time Frame: change from T0 (entry to study) at post-treatment (2-4 weeks after T0), change from T0 at 4 weeks follow-up (6-8 weeks after T0)
10 Meter Walk Test (10mWT) | Time Frame: change from T0 (entry to study) at post-treatment (2-4 weeks after T0), change from T0 at 4 weeks follow-up (6-8 weeks after T0)
6 Minute Walk Test (6MWT) | Time Frame: change from T0 (entry to study) at post-treatment (2-4 weeks after T0), change from T0 at 4 weeks follow-up (6-8 weeks after T0)
Weekly diary | Time Frame: change from T0 (baseline), at week 1 - 8 (1 - 8 week after T0)
  Participants will also be asked to complete a weekly diary. Each week, participants will be prompted to document circumstances in their daily life that either prevented or instead supported engaging in PA in an open-ended questionnaire. More specifically, participants will be asked to answer the following questions:
  * What kind of goals in terms of PA did you pursue this week?
  * What prevented you this week from engaging in physical activities?
  * What facilitated this week engaging in physical activities?
  * What would have been helpful to increase PA?
  * What was your experience with the activity trackers this week?

CONTACTS AND LOCATIONS:
Overall Officials: Viktor von Wyl, Prof. Dr., Principal Investigator — University of Zurich
Locations (1):
- Kliniken Valens, Valens, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chiu C, Bishop M, Pionke JJ, Strauser D, Santens RL. Barriers to the Accessibility and Continuity of Health-Care Services in People with Multiple Sclerosis: A Literature Review. Int J MS Care. 2017 Nov-Dec;19(6):313-321. doi: 10.7224/1537-2073.2016-016. PMID 29270089
- [Background] Block VJ, Bove R, Zhao C, Garcha P, Graves J, Romeo AR, Green AJ, Allen DD, Hollenbach JA, Olgin JE, Marcus GM, Pletcher MJ, Cree BAC, Gelfand JM. Association of Continuous Assessment of Step Count by Remote Monitoring With Disability Progression Among Adults With Multiple Sclerosis. JAMA Netw Open. 2019 Mar 1;2(3):e190570. doi: 10.1001/jamanetworkopen.2019.0570. PMID 30874777
- [Background] Heine M, van de Port I, Rietberg MB, van Wegen EE, Kwakkel G. Exercise therapy for fatigue in multiple sclerosis. Cochrane Database Syst Rev. 2015 Sep 11;2015(9):CD009956. doi: 10.1002/14651858.CD009956.pub2. PMID 26358158
- [Background] Motl RW, McAuley E, Snook EM. Physical activity and multiple sclerosis: a meta-analysis. Mult Scler. 2005 Aug;11(4):459-63. doi: 10.1191/1352458505ms1188oa. PMID 16042230